CLINICAL TRIAL: NCT00394433
Title: A Phase II Trial of Docetaxel, Cisplatin, Irinotecan and Bevacizumab (TPCA) in Metastatic Esophageal and Gastric Cancer
Brief Title: Docetaxel, Cisplatin, Irinotecan and Bevacizumab (TPCA) in Metastatic Esophageal and Gastric Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Brigham and Women's Hospital (Other); Massachusetts General Hospital (Other); Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, Peter C. Enzinger, MD, Overall PI, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06-100
Record Dates: First submitted 2006-10-31; First posted 2006-11-01 (Estimated); Results first posted 2017-01-16 (Estimated); Last update posted 2017-08-01 (Actual); Status verified 2017-07

CONDITIONS: Esophageal Cancer; Stomach Cancer
Keywords: TPCA; Taxotere; Platinum; Avastin; Camptosar; gastric cancer
MeSH Terms: conditions — Esophageal Neoplasms; Stomach Neoplasms | interventions — Bevacizumab; Docetaxel; Cisplatin; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Docetaxel, Cisplatin, Irinotecan and Bevacizumab (TPCA) (Experimental): Patients received bevacizumab 10 mg/kg IV on day 1 every 3 weeks while on study. Additionally, they received docetaxel 30 mg/m2 IV over 30 minutes, followed by cisplatin 25 mg/m2 IV over 30 minutes, followed by irinotecan 50 mg/m2 IV over 30 minutes on days 1 and 8 of each 3-week cycle until disease progression or unacceptable toxicity. Dose reductions were not permitted for bevacizumab although treatment could be held up to 2 months. If bevacizumab was discontinued, treatment with other agents could continue. When docetaxel, cisplatin, or irinotecan was held on day 1 of a cycle, all agents were held.
  Interventions: Drug: Bevacizumab; Drug: Docetaxel; Drug: Cisplatin; Drug: Irinotecan

INTERVENTIONS:
Drug: Bevacizumab
  Other Names: Avastin
Drug: Docetaxel
  Other Names: Taxotere, Docefrez
Drug: Cisplatin
  Other Names: Platinol-AQ, Platinol
Drug: Irinotecan
  Other Names: Camptosar

SUMMARY:
The purpose of this research study is to determine if the combination of docetaxel, cisplatin, irinotecan and bevacizumab will help shrink metastatic esophageal or gastric cancer and how the cancer responds to this combination. Bevacizumab is a new drug that is believed to stop the formation of new blood vessels that carry nutrients to tumors. Bevacizumab is approved for use in metastatic colon and rectal cancer. Docetaxel, cisplatin and irinotecan are traditional chemotherapy agents that have been tested together in another clinical trial for esophageal and gastric cancer. It is hoped that adding bevacizumab to this regimen will make the treatment more effective.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

To determine the 10-month progression-free survival rate for the combination of TPC and Bevacizumab in patients with metastatic esophageal or gastric cancer

Secondary

* To determine the response rate (RECIST) and median duration of response
* To determine overall survival
* To determine toxicity

Exploratory

* To explore if 7/7 and 7/6 UGT1A1 polymorphisms correlate with grade III/IV irinotecan-related diarrhea and neutropenia when irinotecan is given at relatively low dose to patients with esophageal and gastric cancer
* To correlate expression of tumoral and serum VEGF with response and survival
* To correlate TGF alpha levels and tumor microvessel density with clinical activity
* To examine circulating endothelial cells (CECs) as surrogate markers of antitumor activity of bevacizumab

DESIGN This trial will use a single stage design to differentiate a >/= 50% rate of 10-month progression-free survival from a </= 30% rate. The proposed regimen would be promising if at least 15 of 35 patients were alive and progression-free at 10 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed, unresectable esophageal or gastric carcinoma (carcinoma=adenocarcinoma or squamous cell carcinoma)
* Measurable disease greater than or equal to 1 cm (longest diameter) by spiral computed tomography (CT) scan or 2 cm or greater by other radiographic technique
* Lesions must be measurable in at least one dimension
* Bone lesions, ascites, and effusions are not measurable
* 18 years of age or older
* ECOG performance status 0 or 1
* Life expectancy of at least 12 weeks
* Adequate bone marrow function
* Adequate renal function
* Adequate liver function

Exclusion Criteria:

* Prior chemotherapy (except as part of pre- or post-operative therapy, completed more than 1 year prior to start day of this protocol)
* History of severe hypersensitivity to bevacizumab, docetaxel, cisplatin, irinotecan, or drugs formulated with polysorbate 80
* Current, recent (within 4 weeks) or planned participation in an experimental drug study
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to Day 0, or anticipation of need for major surgical procedure during the course of the study
* Minor surgical procedures, such as fine needle aspirations, port-a-cath placement, or core biopsies within 7 days prior to Day 0 of study
* Myocardial infarction or stroke in past 6 months
* Blood pressure of > 150/100 mmHg
* Unstable angina
* New York Heart Association (NYHA) grade II or greater congestive heart failure
* Clinically significant peripheral vascular disease
* Persistent bleeding from primary tumor, while off anticoagulants, requiring repeated transfusions
* Evidence of bleeding diathesis or coagulopathy
* Uncontrolled serious medical or psychiatric illness
* Uncontrolled diarrhea
* Peripheral neuropathy > grade 1
* Clinically apparent central nervous system metastases or carcinomatous meningitis
* Other active malignancy other than non-melanoma skin cancer or in situ cervical carcinoma.
* Urine protein: creatinine ratio of 1.0 or greater at screening
* History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months prior to Day 1
* Serious non-healing wound, ulcer, or bone fracture
* Pregnant or breast-feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2006-09; Primary Completion 2008-11 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Enzinger, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (3):
- United States (3):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients (n=38) were enrolled between September 2006 and March 2008.
Period: Overall Study
Arm/Group | Docetaxel, Cisplatin, Irinotecan and Bevacizumab (TPCA)
Started | 38
Evaluable and Treated | 35
Completed | 35
Not Completed | 3
Not completed — Adverse Event | 2
Not completed — Alternative Therapy | 1

BASELINE CHARACTERISTICS:
Population: The analysis dataset is comprised of all enrolled patients.
Arm/Group | Docetaxel, Cisplatin, Irinotecan and Bevacizumab (TPCA)
Number analyzed (Participants) | 38
Age, Continuous [Median (Full Range); unit: years] | 58 [31 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 32
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 33
  Black or African American | 2
  Hispanic | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 38
Primary Site of Disease [Count of Participants; unit: Participants]
  Esophageal | 13
  Gastroesophageal junction | 9
  Gastric | 16

OUTCOME MEASURES:

1. Primary Outcome: 10-month Progression-Free Survival Rate
Description: 10-month progression-free survival rate is the probability of patients remaining alive and progression-free at 10-months from study entry estimated using Kaplan-Meier methods. Per RECIST 1.0 criteria: progressive disease (PD) is at least a 20% increase in the sum of longest diameter (LD) of target lesions taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions. PD for the evaluation of non-target lesions is the appearance of one or more new lesions and/or unequivocal progression of non-target lesions.
Time Frame: Disease was evaluated radiologically at baseline and every 2 cycles on treatment; Treatment continued until disease progression or unacceptable toxicity. Relevant for this endpoint was disease status at 10 months.
Population: The analysis dataset is comprised of all enrolled patients.
Measure: Number (95% Confidence Interval); unit: probability (%)
Arm/Group | Docetaxel, Cisplatin, Irinotecan and Bevacizumab (TPCA)
Number analyzed (Participants) | 38
probability (%) | 40.0 [21.5 to 55.1]

2. Secondary Outcome: Best Response
Description: Best response on treatment was based on RECIST 1.0 criteria: Complete Response (CR) is complete disappearance of all target lesions; Partial Response (PR) is at least a 30% decrease in the sum of longest diameter (LD) of target lesions, taking as reference baseline sum LD. Both require confirmation no fewer than 4 weeks apart. CR/PR assumes at a minimum incomplete response/stable disease (SD) for the evaluation of non-target lesions and absence of new lesions. Progressive disease (PD) is at least a 20% increase in the sum of longest diameter of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions. PD for the evaluation of non-target lesions is the appearance of one or more new lesions and/or unequivocal progression of non-target lesions. Stable disease is defined as any condition not meeting above criteria.
Time Frame: Disease was evaluated radiologically at baseline and every 2 cycles on treatment. Treatment continued until disease progression or unacceptable toxicity. Treatment duration was a median of 6 cycles/18 weeks given 3-week cycle length (range 1-26 cycles).
Population: The analysis dataset is comprised of all treated and evaluable patients.
Measure: Number; unit: participants
Arm/Group | Docetaxel, Cisplatin, Irinotecan and Bevacizumab (TPCA)
Number analyzed (Participants) | 35
participants
  Partial Response | 23
  Stable Disease | 7
  Progressive Disease | 5

3. Secondary Outcome: Overall Survival
Description: Overall survival is defined as the time from study entry to death or date last known alive and estimate using Kaplan-Meier (KM) methods.
Time Frame: Patients in the study cohort were followed for a median of 12.2 month (up to 40 months).
Population: The analysis dataset is comprised of all enrolled patients.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Docetaxel, Cisplatin, Irinotecan and Bevacizumab (TPCA)
Number analyzed (Participants) | 38
months | 14.9 [9.6 to 18.4]

4. Secondary Outcome: Progression-Free Survival
Description: Progression-free survival based on the Kaplan-Meier method is defined as the duration of time from study entry to documented disease progression (PD) requiring removal from the study or death. Patients alive and progression-free at last follow-up are censored. Per RECIST 1.0 criteria: progressive disease is at least a 20% increase in the sum of longest diameter (LD) of target lesions taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions. PD for the evaluation of non-target lesions is the appearance of one or more new lesions and/or unequivocal progression of non-target lesions.
Time Frame: as for outcome 2
Population: The analysis dataset is comprised of all enrolled patients.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Docetaxel, Cisplatin, Irinotecan and Bevacizumab (TPCA)
Number analyzed (Participants) | 38
months | 8.9 [5.4 to 10.3]

ADVERSE EVENTS:
Time Frame: Adverse events were assessed weeks 1 and 2 each cycle throughout treatment. Treatment continued until disease progression or unacceptable toxicity. Treatment duration was a median of 6 cycles/18 weeks given 3-week cycle length (range 1-26 cycles).
Description: Maximum grade toxicity by type was first calculated. Serious AEs were defined as events with treatment-attribution of possibly, probably or definitely and grade 3 or higher per CTCAEv3. Other AEs were defined as events with treatment-attribution of possible, probable or definite and grades 1 or 2 per CTCAEv3. No further data is available to specify classification of other beyond the general term.
Arm/Group | Docetaxel, Cisplatin, Irinotecan and Bevacizumab (TPCA)
Serious Adverse Events (participants affected / at risk) | 30/38
Other Adverse Events (participants affected / at risk) | 37/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Docetaxel, Cisplatin, Irinotecan and Bevacizumab (TPCA) (N=38)
Hemoglobin (Blood and lymphatic system disorders) | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 6
Constipation (Gastrointestinal disorders) | 1
Diarrhea w/o prior colostomy (Gastrointestinal disorders) | 16
Dysphagia (Gastrointestinal disorders) | 1
Esophagitis (Gastrointestinal disorders) | 2
Ileus (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 4
Vomiting (Gastrointestinal disorders) | 2
Upper GI, hemorrhage NOS (Gastrointestinal disorders) | 2
Abdomen, pain (Gastrointestinal disorders) | 2
Fatigue (General disorders) | 7
Allergic reaction (Immune system disorders) | 1
Infection w/ gr3-4 neut, vulva (Infections and infestations) | 1
Infection Gr0-2 neut, lung (Infections and infestations) | 1
Infection Gr 0-2 neut, blood (Infections and infestations) | 1
Leukocytes (Investigations) | 9
Lymphopenia (Investigations) | 12
Neutrophils (Investigations) | 12
Weight gain (Investigations) | 1
INR (Investigations) | 1
ALT, SGPT (Investigations) | 1
Anorexia (Metabolism and nutrition disorders) | 6
Dehydration (Metabolism and nutrition disorders) | 5
Hypoalbuminemia (Metabolism and nutrition disorders) | 1
Hypocalcemia (Metabolism and nutrition disorders) | 3
Hyperglycemia (Metabolism and nutrition disorders) | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 2
Hypophosphatemia (Metabolism and nutrition disorders) | 2
Hypokalemia (Metabolism and nutrition disorders) | 6
Hyponatremia (Metabolism and nutrition disorders) | 4
Neuropathy-motor (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Hiccoughs (Respiratory, thoracic and mediastinal disorders) | 1
Nasal cavity/paranasal sinus reaction (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary/Upper Respiratory-other (Respiratory, thoracic and mediastinal disorders) | 1
Hypertension (Vascular disorders) | 2
Hypotension (Vascular disorders) | 1
Thrombosis/thrombus/embolism (Vascular disorders) | 6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Docetaxel, Cisplatin, Irinotecan and Bevacizumab (TPCA) (N=38)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 3
Hemorrhage (Vascular disorders) | 1
Hemoglobin (Blood and lymphatic system disorders) | 28
Hematologic (Blood and lymphatic system disorders) | 5
Lymphatics (Blood and lymphatic system disorders) | 1
Hearing (Ear and labyrinth disorders) | 1
External ear, pain (Ear and labyrinth disorders) | 1
Vision-blurred (Eye disorders) | 1
Tearing (Eye disorders) | 3
Ocular (Eye disorders) | 1
Ascites (non-malignant) (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 22
Diarrhea w/o prior colostomy (Gastrointestinal disorders) | 19
Distention/bloating, abdominal (Gastrointestinal disorders) | 3
Dry mouth (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 4
Flatulence (Gastrointestinal disorders) | 7
Dyspepsia (Gastrointestinal disorders) | 7
Hemorrhoids (Gastrointestinal disorders) | 1
Muco/stomatitis by exam, oral cavity (Gastrointestinal disorders) | 7
Muco/stomatitis (symptom) oral cavity (Gastrointestinal disorders) | 3
Nausea (Gastrointestinal disorders) | 30
Ulcer, rectum (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 24
GI-other (Gastrointestinal disorders) | 8
Rectum, hemorrhage (Gastrointestinal disorders) | 1
Abdomen, pain (Gastrointestinal disorders) | 18
Esophagus, pain (Gastrointestinal disorders) | 1
Oral cavity, pain (Gastrointestinal disorders) | 2
Rectum, pain (Gastrointestinal disorders) | 1
Stomach, pain (Gastrointestinal disorders) | 7
Fatigue (General disorders) | 28
Fever w/o neutropenia (General disorders) | 6
Rigors/chills (General disorders) | 4
Constitutional (General disorders) | 1
Injection site reaction (General disorders) | 1
Edema limb (General disorders) | 5
Chest/thoracic pain NOS (General disorders) | 5
Pain NOS (General disorders) | 3
Pain-other (General disorders) | 3
Liver, pain (Hepatobiliary disorders) | 1
Allergic reaction (Immune system disorders) | 2
Allergy-other (Immune system disorders) | 1
Infection w/ gr3-4 neut, skin (Infections and infestations) | 1
Infection Gr0-2 neut, lung (Infections and infestations) | 1
Infection-other (Infections and infestations) | 2
Wound - non-infectious (Injury, poisoning and procedural complications) | 2
Leukocytes (Investigations) | 20
Lymphopenia (Investigations) | 7
Neutrophils (Investigations) | 11
Platelets (Investigations) | 8
Weight gain (Investigations) | 1
Weight loss (Investigations) | 7
Alkaline phosphatase (Investigations) | 7
ALT, SGPT (Investigations) | 8
AST, SGOT (Investigations) | 8
Bilirubin (Investigations) | 2
Creatinine (Investigations) | 6
Anorexia (Metabolism and nutrition disorders) | 18
Dehydration (Metabolism and nutrition disorders) | 15
Hypoalbuminemia (Metabolism and nutrition disorders) | 13
Bicarbonate (Metabolism and nutrition disorders) | 8
Hypocalcemia (Metabolism and nutrition disorders) | 15
Hyperglycemia (Metabolism and nutrition disorders) | 13
Hypoglycemia (Metabolism and nutrition disorders) | 2
Hypomagnesemia (Metabolism and nutrition disorders) | 10
Hypophosphatemia (Metabolism and nutrition disorders) | 3
Hyperkalemia (Metabolism and nutrition disorders) | 10
Hypokalemia (Metabolism and nutrition disorders) | 6
Hypernatremia (Metabolism and nutrition disorders) | 2
Hyponatremia (Metabolism and nutrition disorders) | 17
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Nonneuropathic lower extr muscle weak (Musculoskeletal and connective tissue disorders) | 1
Nonneuropathic generalized weakness (Musculoskeletal and connective tissue disorders) | 7
Back, pain (Musculoskeletal and connective tissue disorders) | 2
Chest wall, pain (Musculoskeletal and connective tissue disorders) | 1
Extremity-limb, pain (Musculoskeletal and connective tissue disorders) | 1
Joint, pain (Musculoskeletal and connective tissue disorders) | 3
Muscle, pain (Musculoskeletal and connective tissue disorders) | 2
Taste disturbance (Nervous system disorders) | 13
Dizziness (Nervous system disorders) | 15
Neuropathy-motor (Nervous system disorders) | 2
Neuropathy-sensory (Nervous system disorders) | 11
Head/headache (Nervous system disorders) | 10
Insomnia (Psychiatric disorders) | 7
Anxiety (Psychiatric disorders) | 3
Depression (Psychiatric disorders) | 3
Libido (Psychiatric disorders) | 1
Glomerular filtration rate (Renal and urinary disorders) | 1
Proteinuria (Renal and urinary disorders) | 1
Urinary frequency/urgency (Renal and urinary disorders) | 1
Pelvic, pain (Reproductive system and breast disorders) | 1
Erectile impotence (Reproductive system and breast disorders) | 1
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 11
Muco/stomatitis (symptom) trachea (Respiratory, thoracic and mediastinal disorders) | 1
Nose, hemorrhage (Respiratory, thoracic and mediastinal disorders) | 13
Throat/pharynx/larynx, pain (Respiratory, thoracic and mediastinal disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 7
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 7
Hiccoughs (Respiratory, thoracic and mediastinal disorders) | 1
Nasal cavity/paranasal sinus reaction (Respiratory, thoracic and mediastinal disorders) | 3
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 1
Voice changes/dysarthria (Respiratory, thoracic and mediastinal disorders) | 12
Pulmonary/Upper Respiratory (Respiratory, thoracic and mediastinal disorders) | 1
Sweating (Skin and subcutaneous tissue disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 2
Alopecia (Skin and subcutaneous tissue disorders) | 19
Nail changes (Skin and subcutaneous tissue disorders) | 4
Pruritus/itching (Skin and subcutaneous tissue disorders) | 1
Rash/desquamation (Skin and subcutaneous tissue disorders) | 2
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 1
Hand-foot reaction (Skin and subcutaneous tissue disorders) | 2
Ulceration (Skin and subcutaneous tissue disorders) | 1
Skin (Skin and subcutaneous tissue disorders) | 5
Petechiae (Skin and subcutaneous tissue disorders) | 1
Scalp, pain (Skin and subcutaneous tissue disorders) | 1
Hypertension (Vascular disorders) | 6
Hypotension (Vascular disorders) | 1
Hot flashes (Vascular disorders) | 3
Hemorrhage (Vascular disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No